CLINICAL TRIAL: NCT00316212
Title: Randomized, Multicenter, Placebo-Controlled, Double-Blind, Parallel Group Study of INS50589 Intravenous Infusion in Subjects Undergoing Coronary Artery Bypass Graft Surgery Involving Cardiopulmonary Bypass
Brief Title: Study of INS50589 Intravenous Infusion in Subjects Undergoing Coronary Artery Bypass Grafting (CABG) Involving Cardiopulmonary Bypass
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 025-102
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Coronary Disease
Keywords: Coronary Artery Bypass Graft Surgery involving Cardiopulmonary Bypass
MeSH Terms: conditions — Coronary Disease

INTERVENTIONS:
Drug: INS50589 Intravenous Infusion

SUMMARY:
The purpose of this trial is to identify a dose or doses of INS50589 intravenous infusion that are well-tolerated and which reduce postoperative bleeding and blood product transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Are scheduled for primary CABG by median sternotomy involving cardiopulmonary bypass
* Willing to receive allogeneic blood product transfusions during and after surgery

Exclusion Criteria:

* Have had previous cardiac surgery
* Have had previous median sternotomy
* Have tendency for bleeding or family history of bleeding
* Have an abnormally low platelet count
* Have received certain anticoagulant or antiplatelet medications within a specified time period prior to the scheduled CABG surgery

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2006-04; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Postoperative chest drainage volume

SECONDARY OUTCOMES:
Requirement for perioperative blood product transfusion
Incidence of complications after surgery

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Baptist Medical Center Princeton, Birmingham, Alabama
  - Cardiology, P.C., Birmingham, Alabama
  - Sharp Memorial Hospital, San Diego, California
  - Memorial Medical Center, Springfield, Illinois
  - St. John's Hospital, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Lutheran Hospital of Indiana, Fort Wayne, Indiana
  - Veterans Affairs Medical Center, Lexington, Kentucky
  - University of Kentucky, Chandler Medical Center, Lexington, Kentucky
  - St. Mary's of Michigan, Saginaw, Michigan
  - Covenant Medical Center, Saginaw, Michigan
  - Viahealth Rochester General Hospital, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Brody School of Medicine, East Carolina University, Greenville, North Carolina
  - Cardiac, Vascular, & Thoracic Surgeons, Inc., Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oklahoma Cardiovascular Associates, Oklahoma City, Oklahoma
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - CardioThoracic Surgery Center, PLC, Jackson, Tennessee
  - Jackson Madison County General Hospital, Jackson, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - The Methodist Hospital, Houston, Texas
  - Winchester Medical Center, Winchester, Virginia
  - FHS Research Center, St. Joseph Medical Center, Tacoma, Washington
  - Northwest Cardiovascular Associates, Tacoma, Washington